CLINICAL TRIAL: NCT04614441
Title: Non-Interventional Collecting Evidences For ILD in Taiwan: Optimized Novel Therapy
Brief Title: NICEFIT-ON: A Study Under Routine Clinical Practice in Taiwan to Observe the Long-term Outcome of People With Certain Types of Lung Disease (PF-ILD, SSc-ILD, IPF) Who Start Treatment With Nintedanib
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0393
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Idiopathic Pulmonary Fibrosis (IPF)
  Interventions: Drug: OFEV®
- Progressive Fibrosing Interstitial Lung Disease (PF-ILD)
  Interventions: Drug: OFEV®
- Systemic Sclerosis-associated-Interstitial Lung Disease (SSc-ILD)
  Interventions: Drug: OFEV®

INTERVENTIONS:
Drug: OFEV® — nintedanib

SUMMARY:
To better understand the clinical characteristics of Idiopathic Pulmonary Fibrosis (IPF) / Systemic Sclerosis-associated-Interstitial Lung Disease (SSc-ILD)/ Progressive Fibrosing Interstitial Lung Disease (PF-ILD) patients treated with nintedanib and biomarkers associated with the disease course, a non-interventional, 3-year, prospective study will be conducted to collect the long-term real-world clinical data on IPF/SSc-ILD/PF-ILD patients newly administered with nintedanib in Taiwan

ELIGIBILITY:
Inclusion Criteria:

This study plans to enroll approximately 500 patients with IPF/SSc-ILD/PF-ILD who newly initiate nintedanib per physicians' discretion within 6 months before participating in the study.

IPF cohort:

* Diagnosed with IPF during the prior 6 months before study enrollment, based on the 2018 ATS/ERS/JRS/ALAT guideline
* Patient ≥ 40 years of age
* Newly initiating nintedanib within 6 months prior to participating in the study
* Providing written informed consent prior to participating in the study
* Having further follow-up possibility with participating physician during the planned study period
* Ability to read and write in local language

SSc-ILD cohort:

* Diagnosed with SSc-ILD during the prior 6 months before study enrollment, based on 2013 ACR/EULAR
* Patient ≥ 20 years of age
* Newly initiating nintedanib OR not receiving nintedanib per physician's discretion (For patients who diagnosed with SSc-ILD but are not treated with nintedanib on physician's discretion, they will apply the same inclusion criteria, with baseline characteristics collected only) within 6 months prior to participating in the study
* Providing written informed consent prior to participating in the study
* Having further follow-up possibility with participating physician during the planned study period
* Ability to read and write in local language

PF-ILD cohort:

* Diagnosed with PF-ILD (PF-ILD patients will be enrolled only after nintedanib acquires the label approval from TFDA) during the prior 6 months before study enrollment. The definition of PF-ILD diagnosis is as follows:

  --Patients who have ILD with a progressive phenotype, but are not diagnosed with IPF, per physician's judgment. The pathophysiology in these patients is characterized by self-sustaining fibrosis and a deterioration in lung function over time, with worsening respiratory symptoms, resistance to immune-modulatory therapies, and ultimately early mortality.
* Patient ≥ 20 years of age
* Newly initiating nintedanib OR not receiving nintedanib per physician's discretion (For patients who diagnosed with PF-ILD but are not treated with nintedanib on physician's discretion, they will apply the same inclusion criteria, with baseline characteristics collected only) within 6 months prior to participating in the study
* Providing written informed consent prior to participating in the study
* Having further follow-up possibility with participating physician during the planned study period
* Ability to read and write in local language

Exclusion Criteria:

- Lung transplantation expected within the next 6 months.

--Included in ongoing interventional trials

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study plans to enroll approximately 500 patients with Idiopathic Pulmonary Fibrosis (IPF) / Systemic Sclerosis-associated-Interstitial Lung Disease (SSc-ILD)/ Progressive Fibrosing Interstitial Lung Disease (PF-ILD) who newly initiate nintedanib per physicians' discretion within 6 months before participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Annual percentage of decline from baseline in Forced Vital Capacity (FVC, %) per cohort of IPF, SSc-ILD, or PF-ILD | Up to 5 years
  IPF: Idiopathic Pulmonary Fibrosis PF-ILD: Progressive Fibrosing Interstitial Lung Disease SSc-ILD: Systemic Sclerosis-associated-Interstitial Lung Disease
Annual decline from baseline in Diffusing capacity of the Lungs for Carbon monoxide (DLco, %) | Up to 5 years
Annual decline from baseline in resting and exercise Oxygen Saturation (SpO2, %) | Up to 5 years

SECONDARY OUTCOMES:
Time to first acute exacerbation (AE) of IPF; or time to ILD worsening for SSc-ILD/PF-ILD after study enrollment | Up to 5 years
Annual change from baseline in St George's Respiratory Questionnaire (SGRQ) for IPF or King's Brief Interstitial Lung (K-BILD) for other ILDs | Up to 5 years
  IPF: Idiopathic Pulmonary Fibrosis ILD: Interstitial Lung Disease
Annual change from baseline in Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) | Up to 5 years
Annual change from baseline in Six-Minutes Walking Test (6MWT) | Up to 5 years
Annual change from baseline in Berlin questionnaire | Up to 5 years
Change from baseline in quantification of biomarkers | Up to 5 years
  Biomarkers include but not limited to Platelet Derived Growth Factor (PDGF), Vascular Endothelial Growth Factor (VEGF), Fibroblast Growth Factor (FGF), Transforming Growth Factor β1 (TGF-β1), Hepatocyte Growth Factor (HGF), Matrix Metalloproteinase (MMP): MMP-1, MMP-7, MMP-9, α-defensin 1, High Mobility Group Box 1 (HMGB1), Tissue of Metalloproteinase (TIMP), Heat-Shock Protein (HSP): HSP-27, bile acid conjugated, Lysophosphatidic Acid (LPA), Lysophosphatidic Acid Receptor 1 (LPAR1), Prostagladin E2 (PGE2), Interleukin (IL): IL-1β, IL-4, IL-18, IL-13, IL-17, Monocyte Chemoattractant Protein 1 (MCP-1), Macrophage Inflammatory Protein 2 (MIP-2), periostin, osteopontin, Surfactant Protein A (SPA), Surfactant Protein D (SPD), Krebs von den Lungen 6 / Mucin 1 (KL-6/MUC1), anti-HSP70 Immunoglobolin (IgG), Bone Morphogenic Protein (BMP), Carbonhydrate Antigen-199 (CA-199), C-Reaktiv Protein degraded by MMPs (CRPM), chemokine ligand (CCL): CCL 2, CCL-18
Mortality (with cause of death): respiratory- and non-respiratory-related death | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (26):
- Taiwan (26):
  - Chang-Hua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital Chiayi, Chiayi City
  - National Taiwan University Hospital-Hsin-Chu Branch, Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Tzu Chi General Hospital, New Taipei City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Cheng Ching Hospital, Taichung
  - Asia University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Cheng Hsin Rehabilitation Medical Center, Taipei
  - Taitung MacKay Memorial Hospital, Taitung
  - TaoYuan General Hospital, Taoyuan
  - Chang Gung Memorial Hospital(Linkou), Taoyuan District
  - National Yang-Ming University Hospital, Yilan
  - National Taiwan University Hospital Yun-Lin Branch, Yunlin County

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
  .
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/